CLINICAL TRIAL: NCT02023112
Title: An Open-label Study to Evaluate the Efficacy and Safety of ABT-450/Ritonavir/ABT-267 (ABT-450/r/ABT-267) Co-administered With Ribavirin (RBV) for 12 or 16 Weeks in Treatment-Naïve and Treatment-Experienced Japanese Adults With Genotype 2 Chronic Hepatitis C Virus (HCV) Infection With and Without Compensated Cirrhosis (GIFT-II)
Brief Title: Study to Evaluate the Efficacy and Safety of ABT-450/Ritonavir/ABT- 267 (ABT-450/r/ABT-267) in Japanese Adults With Genotype 2 Chronic Hepatitis C Virus (HCV) Infection
Acronym: GIFT-II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M14-153
Record Dates: First submitted 2013-12-23; First posted 2013-12-30 (Estimated); Results first posted 2016-05-13 (Estimated); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Hepatitis C Virus
Keywords: Japanese; Hepatitis C; Treatment naive; Treatment experienced; Genotype 2; Ombitasvir; Paritaprevir; Ritonavir; Ribavirin; VIEKIRAX Combination Tablets
MeSH Terms: conditions — Hepatitis C | interventions — ombitasvir; paritaprevir; Ritonavir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABT-450/r/ABT-267 plus RBV for 12 weeks (Experimental): ABT-450/r/ABT-267 (150/100/25 mg once daily) plus weight-based ribavirin (RBV; 400 to 1,000 mg/day, divided twice daily) for 12 weeks
  Interventions: Drug: ABT-450/r/ABT-267; Drug: Ribavirin
- ABT-450/r/ABT-267 plus RBV for 16 weeks (Experimental): ABT-450/r/ABT-267 (150/100/25 mg once daily) plus weight-based RBV (400 to 1,000 mg/day, divided twice daily) for 16 weeks
  Interventions: Drug: ABT-450/r/ABT-267; Drug: Ribavirin

INTERVENTIONS:
Drug: ABT-450/r/ABT-267 — Tablet; ABT-450 coformulated with ritonavir and ABT-267
  Other Names: ABT-267 also known as ombitasvir; ABT-450 also known as paritaprevir; ritonavir also known as Norvir; VIEKIRAX Combination Tablets; VIEKIRA Combination Tablets; Technivie; Qurevo
Drug: Ribavirin — Capsule

SUMMARY:
This is a Phase 3, randomized, open-label, multicenter study, enrolling non-cirrhotic and cirrhotic subjects. The purpose of this study is to evaluate the efficacy and safety of ABT-450/r/ABT-267 co-administered with weight-based RBV for 12 or 16 weeks in adult chronic HCV genotype 2-infected treatment-naïve and interferon (IFN) treatment-experienced subjects with and without compensated cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV-infection prior to study enrollment
* Screening laboratory result indicating HCV genotype 2 infection
* Subject has plasma HCV ribonucleic acid (RNA) level greater than 10,000 IU/mL at Screening
* Voluntarily sign an informed consent

Exclusion Criteria:

* Co-infection of Hepatitis B Virus (HBV), human immunodeficiency virus (HIV) and any HCV genotype other than genotype 2
* Prior therapy with direct acting antiviral agents for the treatment of HCV, including telaprevir, simeprevir and boceprevir
* Any cause of liver disease other than chronic HCV-infection, including but not limited to the following: hemochromatosis; alpha-1 antitrypsin deficiency; Wilson's disease; autoimmune hepatitis; alcoholic liver disease; drug-related liver disease
* Clinically significant laboratory abnormalities
* Uncontrolled clinically significant disease, disorder or medical illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yasunori Yachi, Study Director — AbbVie

REFERENCES:
- [Background] Sato K, Chayama K, Alves K, Toyoda H, Suzuki F, Kato K, Rodrigues L Jr, Zhang X, Setze C, Pilot-Matias T, Burroughs M, Redman R, Kumada H. Randomized Phase 3 Trial of Ombitasvir/Paritaprevir/Ritonavir and Ribavirin for Hepatitis C Virus Genotype 2-Infected Japanese Patients. Adv Ther. 2017 Jun;34(6):1449-1465. doi: 10.1007/s12325-017-0506-y. Epub 2017 May 23. PMID 28536999

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ABT-450/r/ABT-267 Plus RBV for 12 Weeks | ABT-450/r/ABT-267 Plus RBV for 16 Weeks
Started | 85 | 86
Completed | 83 | 85
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- ABT-450/r/ABT-267 Plus RBV for 12 Weeks: ABT-450/r/ABT-267 (150/100/25 mg once daily) plus weight-based RBV (400 to 1,000 mg/day, divided twice daily) for 12 weeks
- Total: Total of all reporting groups
Arm/Group | ABT-450/r/ABT-267 Plus RBV for 12 Weeks | ABT-450/r/ABT-267 Plus RBV for 16 Weeks | Total
Number analyzed (Participants) | 85 | 86 | 171
Age, Customized [Number; unit: participants]
  < 65 years | 56 | 62 | 118
  ≥ 65 years | 29 | 24 | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 48 | 88
  Male | 45 | 38 | 83

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Non-cirrhotic, Treatment-naive Participants in Each Treatment Group With a Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: The percentage of participants with sustained virologic response (plasma Hepatitis C virus ribonucleic acid [HCV RNA] level less than the lower limit of quantitation [< LLOQ]) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after last dose of study drug
Population: Primary efficacy population: all treatment-naïve, noncirrhotic participants in the intent-to-treat (ITT) population (all randomized participants who received at least 1 dose of study drug).
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r/ABT-267 Plus RBV for 12 Weeks | ABT-450/r/ABT-267 Plus RBV for 16 Weeks
Number analyzed (Participants) | 48 | 47
percentage of participants | 75.0 | 91.5
Statistical Analysis 1: Comparison: ABT-450/r/ABT-267 Plus RBV for 16 Weeks; Among non-cirrhotic treatment-naïve participants, superiority of the 16-week treatment arm to a clinically relevant threshold. Lower bound of 95% confidence interval (LCB) must have exceeded 67% to achieve superiority. Threshold indicates value the LCB had to exceed to demonstrate superiority for the treatment arm and was based on the SVR rates with pegylated-interferon (IFN) alfa-2a or 2b/RBV in treatment-naïve, noncirrhotic HCV genotype 2-infected participants; Test type: Superiority or Other; percentage of participants with SVR12 = 91.5, 95% CI 2-sided [80.1 to 96.6] — Tested using the following hierarchical order: among non-cirrhotic treatment-naïve participants 1) superiority of 16-week treatment arm to a clinically relevant threshold; 2) superiority of 12-week treatment arm to a clinically relevant threshold
Statistical Analysis 2: Comparison: ABT-450/r/ABT-267 Plus RBV for 12 Weeks; Among non-cirrhotic treatment-naïve participants, superiority of the 12-week treatment arm to a clinically relevant threshold. LCB must have exceeded 67% to achieve superiority. Threshold indicates value the LCB had to exceed to demonstrate superiority for the treatment arm and was based on the SVR rates with pegylated-IFN alfa-2a or 2b/RBV in treatment-naïve, noncirrhotic HCV genotype 2-infected participants; Test type: Superiority or Other; percentage of participants with SVR12 = 75.0, 95% CI 2-sided [61.2 to 85.1] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Percentage of Participants in Each Treatment Arm With On-treatment Virologic Failure During the Treatment Period
Description: On-treatment virologic failure was defined as rebound (confirmed HCV RNA ≥ LLOQ after HCV RNA < LLOQ during treatment, or confirmed increase from nadir in HCV RNA [> 1 log10 IU/mL above nadir] at any time point during treatment) or failure to suppress HCV during treatment (all on-treatment values of HCV RNA ≥ LLOQ with at least 6 weeks of treatment).
Time Frame: 12 or 16 weeks (end of treatment period)
Population: Primary efficacy population: all treatment-naïve, noncirrhotic participants in the ITT population (all randomized participants who received at least 1 dose of study drug).
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r/ABT-267 Plus RBV for 12 Weeks | ABT-450/r/ABT-267 Plus RBV for 16 Weeks
Number analyzed (Participants) | 48 | 47
percentage of participants
  Overall | 8.3 | 8.5
  Rebound | 8.3 | 8.5
  Failure to suppress | 0 | 0

3. Secondary Outcome: Percentage of Participants With Post-treatment Relapse
Description: Relapse by post-treatment Week 12 was defined as confirmed HCV RNA ≥ LLOQ between end of treatment and 12 weeks after last actual dose of study drug for a participant with HCV RNA < LLOQ at the final treatment visit and who completed study treatment. Completion of treatment was defined as a study drug duration ≥ 77 days for the 12-week treatment arm or ≥ 105 days for the 16-week treatment arm.
Time Frame: within 12 weeks after the last dose of study drug
Population: Primary efficacy population: all treatment-naïve, noncirrhotic participants in the ITT population (all randomized participants who received at least 1 dose of study drug) with HCV RNA < LLOQ at the final treatment visit who completed treatment.
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r/ABT-267 Plus RBV for 12 Weeks | ABT-450/r/ABT-267 Plus RBV for 16 Weeks
Number analyzed (Participants) | 41 | 47
percentage of participants | 12.2 | 0

4. Secondary Outcome: Percentage of Participants With SVR12 Weeks Post-treatment for Each Treatment Arm Within Different Subpopulations
Description: The percentage of participants with SVR12 in each treatment arm within the following subpopulations: noncirrhotic participants; noncirrhotic treatment-experienced (T-exp) participants; noncirrhotic participants who relapsed after prior IFN-based therapy (relapsers); noncirrhotic T-exp participants who were non-responders to prior IFN-based therapy; noncirrhotic T-exp participants who were intolerant to IFN-based therapy; participants with compensated cirrhosis.
Time Frame: 12 weeks after last dose of study drug
Population: ITT population: all randomized participants who received at least 1 dose of study drug; n=participants in given subpopulation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-450/r/ABT-267 Plus RBV for 12 Weeks | ABT-450/r/ABT-267 Plus RBV for 16 Weeks
Number analyzed (Participants) | 85 | 86
percentage of participants
  All participants; n=85, 86 | 72.9 [62.7 to 81.2] | 81.4 [71.9 to 88.2]
  Noncirrhotic participants; n=80, 80 | 72.5 [61.9 to 81.1] | 85.0 [75.6 to 91.2]
  Noncirrhotic T-exp; n=32, 33 | 68.8 [51.4 to 82.0] | 75.8 [59.0 to 87.2]
  Noncirrhotic T-exp Relapser; n=15, 16 | 80.0 [54.8 to 93.0] | 93.8 [71.7 to 98.9]
  Noncirrhotic T-exp Nonresponder; n=5, 6 | 40.0 [11.8 to 76.9] | 50.0 [18.8 to 81.2]
  Noncirrhotic T-exp IFN-intolerant; n=12, 11 | 66.7 [39.1 to 86.2] | 63.6 [35.4 to 84.8]
  Cirrhotic Participants; n=5, 6 | 80.0 [37.6 to 96.4] | 33.3 [9.7 to 70.0]

5. Secondary Outcome: Percentage of Participants in Each Treatment Arm With On-treatment Virologic Failure During the Treatment Period for Each Treatment Arm Within Different Subpopulations
Description: The percentage of participants with on-treatment virologic failure in each treatment arm within the following subpopulations: noncirrhotic participants; noncirrhotic treatment-experienced (T-exp) participants; participants with compensated cirrhosis.
  On-treatment virologic failure was defined as rebound (confirmed HCV RNA ≥ LLOQ after HCV RNA < LLOQ during treatment, or confirmed increase from nadir in HCV RNA [> 1 log10 IU/mL above nadir] at any time point during treatment) or failure to suppress HCV during treatment (all on-treatment values of HCV RNA ≥ LLOQ with at least 6 weeks of treatment).
Time Frame: 12 or 16 weeks (end of treatment period)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r/ABT-267 Plus RBV for 12 Weeks | ABT-450/r/ABT-267 Plus RBV for 16 Weeks
Number analyzed (Participants) | 85 | 86
percentage of participants
  All Participants: Overall; n=85, 86 | 15.3 | 16.3
  All Participants: Rebound; n=85, 86 | 15.3 | 15.1
  All Participants: Failure to Suppress; n=85, 86 | 4.7 | 4.7
  Noncirrhotic: Overall; n=80, 80 | 15.0 | 13.8
  Noncirrhotic: Rebound; n=80, 80 | 15.0 | 12.5
  Noncirrhotic: Failure to Suppress; n=80, 80 | 3.8 | 3.8
  Noncirrhotic T-exp: Overall; n=32, 33 | 25.0 | 21.2
  Noncirrhotic T-exp: Rebound; n=32, 33 | 25.0 | 18.2
  Noncirrhotic T-exp: Failure to Suppress; n=32, 33 | 9.4 | 9.1
  Cirrhotic: Overall; n=5, 6 | 20.0 | 50.0
  Cirrhotic: Rebound; n=5, 6 | 20.0 | 50.0
  Cirrhotic: Failure to Suppress; n=5, 6 | 20.0 | 16.7

6. Secondary Outcome: Percentage of Participants With Post-treatment Relapse Within Different Subpopulations
Description: The percentage of participants with relapse by post-treatment Week 12 in each treatment arm within the following subpopulations: noncirrhotic participants; noncirrhotic treatment-experienced (T-exp) participants; participants with compensated cirrhosis.
  Relapse by post-treatment Week 12 was defined as confirmed HCV RNA ≥ LLOQ between end of treatment and 12 weeks after last actual dose of study drug for a participant with HCV RNA < LLOQ at the final treatment visit and who completed study treatment. Completion of treatment was defined as a study drug duration ≥ 77 days for the 12-week treatment arm or ≥ 105 days for the 16-week treatment arm.
Time Frame: within 12 weeks after the last dose of study drug
Population: ITT population: all randomized participants who received at least 1 dose of study drug with HCV RNA < LLOQ at the final treatment visit who completed treatment; n=participants in given subpopulation.
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r/ABT-267 Plus RBV for 12 Weeks | ABT-450/r/ABT-267 Plus RBV for 16 Weeks
Number analyzed (Participants) | 69 | 70
percentage of participants
  All Participants; n=69, 70 | 10.1 | 0
  Noncirrhotic Participants; n=65, 68 | 10.8 | 0
  Noncirrhotic T-exp Participants; n=24, 25 | 8.3 | 0
  Cirrhotic Participants; n=4, 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: Non-serious adverse events collected from initiation of study drug through 30 days post-study drug dosing (12 weeks or 16 weeks, depending on arm assignment); serious adverse events collected from signing of Informed Consent up to Post-treatment Week 48.
Groups:
- ABT-450/r/ABT-267 Plus RBV for 12 Weeks (Non-cirrhotic): ABT-450/r/ABT-267 (150/100/25 mg once daily) plus weight-based RBV (400 to 1,000 mg/day, divided twice daily) for 12 weeks in non-cirrhotic participants
- ABT-450/r/ABT-267 Plus RBV for 16 Weeks (Non-cirrhotic): ABT-450/r/ABT-267 (150/100/25 mg once daily) plus weight-based RBV (400 to 1,000 mg/day, divided twice daily) for 16 weeks in non-cirrhotic participants
- ABT-450/r/ABT-267 Plus RBV for 12 Weeks (Cirrhotic): ABT-450/r/ABT-267 (150/100/25 mg once daily) plus weight-based RBV (400 to 1,000 mg/day, divided twice daily) for 12 weeks in cirrhotic participants
- ABT-450/r/ABT-267 Plus RBV for 16 Weeks (Cirrhotic): ABT-450/r/ABT-267 (150/100/25 mg once daily) plus weight-based RBV (400 to 1,000 mg/day, divided twice daily) for 16 weeks in cirrhotic participants
Arm/Group | ABT-450/r/ABT-267 Plus RBV for 12 Weeks (Non-cirrhotic) | ABT-450/r/ABT-267 Plus RBV for 16 Weeks (Non-cirrhotic) | ABT-450/r/ABT-267 Plus RBV for 12 Weeks (Cirrhotic) | ABT-450/r/ABT-267 Plus RBV for 16 Weeks (Cirrhotic)
Serious Adverse Events (participants affected / at risk) | 0/80 | 3/80 | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 52/80 | 53/80 | 3/5 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-450/r/ABT-267 Plus RBV for 12 Weeks (Non-cirrhotic) (N=80) | ABT-450/r/ABT-267 Plus RBV for 16 Weeks (Non-cirrhotic) (N=80) | ABT-450/r/ABT-267 Plus RBV for 12 Weeks (Cirrhotic) (N=5) | ABT-450/r/ABT-267 Plus RBV for 16 Weeks (Cirrhotic) (N=6)
GASTRITIS ALCOHOLIC (Gastrointestinal disorders) | 0 | 1 | 0 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 0 | 1 | 0 | 0
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-450/r/ABT-267 Plus RBV for 12 Weeks (Non-cirrhotic) (N=80) | ABT-450/r/ABT-267 Plus RBV for 16 Weeks (Non-cirrhotic) (N=80) | ABT-450/r/ABT-267 Plus RBV for 12 Weeks (Cirrhotic) (N=5) | ABT-450/r/ABT-267 Plus RBV for 16 Weeks (Cirrhotic) (N=6)
ANAEMIA (Blood and lymphatic system disorders) | 16 | 20 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 4 | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 5 | 3 | 0 | 0
FATIGUE (General disorders) | 6 | 2 | 0 | 0
MALAISE (General disorders) | 4 | 7 | 0 | 0
PYREXIA (General disorders) | 2 | 4 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 10 | 13 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 4 | 0 | 0
BLOOD BILIRUBIN INCREASED (Investigations) | 16 | 14 | 0 | 1
BLOOD CHOLESTEROL DECREASED (Investigations) | 3 | 4 | 0 | 0
HAEMOGLOBIN DECREASED (Investigations) | 6 | 4 | 1 | 0
NEUTROPHIL COUNT DECREASED (Investigations) | 1 | 4 | 0 | 0
RED BLOOD CELL COUNT DECREASED (Investigations) | 4 | 3 | 0 | 0
RETICULOCYTE COUNT INCREASED (Investigations) | 6 | 5 | 0 | 0
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 | 4 | 0 | 0
HEADACHE (Nervous system disorders) | 11 | 6 | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 7 | 9 | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 4 | 4 | 0 | 0
HEAT ILLNESS (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
BLOOD URIC ACID INCREASED (Investigations) | 0 | 0 | 1 | 0
DIZZINESS (Nervous system disorders) | 2 | 2 | 0 | 1
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
PALPITATIONS (Cardiac disorders) | 1 | 0 | 0 | 1
VITREOUS HAEMORRHAGE (Eye disorders) | 0 | 0 | 0 | 1
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
SOMNOLENCE (Nervous system disorders) | 0 | 0 | 1 | 0
POLLAKIURIA (Renal and urinary disorders) | 0 | 0 | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 0 | 0 | 1 | 0
HOT FLUSH (Vascular disorders) | 0 | 1 | 1 | 0
HYPOTENSION (Vascular disorders) | 2 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.